CLINICAL TRIAL: NCT06364631
Title: First Line Randomised Study Platform to Optimize Treatment in Patients With Metastatic Renal Cell Carcinoma
Brief Title: CARE1 Pragmatic Clinical Trial
Acronym: CARE1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: European Commission (Other); CRIS Cancer Foundation (Unknown); National Cancer Institute, France (Other Government); Rennes University Hospital (Other); University Hospital, Essen (Other); Fundació Privada Institut d'Investigació Oncològica de Vall d'Hebron (Unknown); The Netherlands Cancer Institute (Other); Servicio Madrileño de Salud, Madrid, Spain (Other); Hospital Universitario 12 de Octubre (Other); Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); Medical University of Vienna (Other); FAKULTNI NEMOCNICE OLOMOUC (Unknown); International Kidney Cancer Coalition (Unknown); Association pour la Recherche sur les Tumeurs du Rein (Unknown); Resilience (Industry); PRIMAA (Unknown); Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-503317-29-00; 2023/3764 (Other: CSET number)
Record Dates: First submitted 2024-04-04; First posted 2024-04-15 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Kidney Cancer; Metastatic Kidney Carcinoma
Keywords: METASTATIC KIDNEY CANCER; METASTATIC KIDNEY CARCINOMA; PRAGMATIC CLINICAL TRIAL; PDL1
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Nivolumab; Ipilimumab; pembrolizumab; cabozantinib; Axitinib; lenvatinib

STUDY DESIGN:
Intervention Model Description: International, multicenter, open-label, randomized, controlled Phase 3 trial - 2 arms (A and B)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: ICI - ICI Combination (Other): Nivolumab (3 mg/kg infusion, every 3 weeks) x 4 doses + ipilimumab (1 mg/kg infusion, every 3 weeks) x 4 doses. At the end of the 4 injections carried out 21 days apart and in the absence of limiting side effects or progression justifying the cessation of the treatment according to the investigating doctor, maintenance treatment with nivolumab will be continued, at a rate of one injection every 2 weeks at a dose of 240 mg or every 4 weeks at a dose of 480 mg depending on the choice of the investigating doctor. Nivolumab will be administered for a maximum of 2 years.
  Patients are required to receive all four doses of NIVO+IPI before beginning NIVO monotherapy except for ipilimumab-induced toxicity compatible with nivolumab maintenance.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- Arm B: VEGFR-TKI- ICI arm (axitinib + pembrolizumab) (Other): Investigator's choice between:
  * Axitinib (5 mg oral twice a day) + pembrolizumab (200 mg flat IV every 3 weeks or 400 mg flat IV every 6 weeks).
  * Cabozantinib (40 mg oral, once a day away from meals) + nivolumab infusion (480 mg flat dose every 4 weeks)
  * Lenvatinib (20 mg oral, once a day) + pembrolizumab (200 mg flat IV every 3 weeks or 400 mg flat IV every 6 weeks)
  Interventions: Drug: Nivolumab; Drug: Pembrolizumab; Drug: Cabozantinib; Drug: Axitinib; Drug: Lenvatinib

INTERVENTIONS:
Drug: Nivolumab — Briefly, nivolumab is administered as an approximately 30-minute (240mg every 2 weeks) or 60-minute (480mg every 4 weeks) IV infusion. Nivolumab is to be administered first. The nivolumab infusion must be promptly followed by a saline flush to clear the line of nivolumab before starting the ipilimumab infusion.
  Other Names: OPDIVO
Drug: Ipilimumab — The second infusion will always be ipilimumab and will start at least 30 minutes after completion of the nivolumab infusion. Ipilimumab is to be administered as an approximately 30-minute IV infusion.
  When administered together, nivolumab and ipilimumab will be administered on Day 1 of each 21-day cycle.
  Other Names: YERVOY
  Arms: Arm A: ICI - ICI Combination
Drug: Pembrolizumab — Pembrolizumab is to be administered as an approximately 30-minute IV infusion.
  Other Names: KEYTRUDA
  Arms: Arm B: VEGFR-TKI- ICI arm (axitinib + pembrolizumab)
Drug: Cabozantinib — Cabozantinib is a medication that is taken orally every day, once a day away from meals at the initial dose of 40 mg/day.
  Other Names: CABOMETYX
  Arms: Arm B: VEGFR-TKI- ICI arm (axitinib + pembrolizumab)
Drug: Axitinib — Axitinib is a medication that is taken orally every day, 2 times a day continuously, at the starting dose of 5mg x2/day.
  Other Names: INLYTA
  Arms: Arm B: VEGFR-TKI- ICI arm (axitinib + pembrolizumab)
Drug: Lenvatinib — Lenvatinib is a medication that is taken orally every day, once a day at the initial dose of 20mg/day.
  Other Names: LENVIMA
  Arms: Arm B: VEGFR-TKI- ICI arm (axitinib + pembrolizumab)

SUMMARY:
Systemic therapy for renal cell carcinoma (RCC) relies on 2 classes of agents: anti-angiogenic targeted therapy (Vascular endothelial growth factor Tyrosine Kinase Inhibitor- VEGFR TKI) and immune checkpoint inhibitor (ICI), targeting either PD1/PDL1 axis or CTLA4. Combination therapy is SOC for clear cell RCC in all guidelines with either ICI-ICI or ICI-VEGFR TKI. However, no head-to-head comparison have been performed between the 2 approaches and patients are treated based on physician decision without clinical /biomarker factors to guide treatment selection. PDL1 staining is, to date, the biomarker that has demonstrated its ability to enrich for overall survival benefit favoring ICI-ICI strategy in PDL1(+) and ICI-VEGFR TKI in PDL1(-) patients.

Study design has been developed to demonstrate that ICI-ICI is superior to ICI-VEGFR TKI in prolonging Overall Survival (OS) for PDL1(+) patients and to demonstrate that ICI-VEGFR TKI is superior to ICI-ICI in prolonging Progression Free Survival (PFS) and OS for PDL1(-) patients.

DETAILED DESCRIPTION:
In 2020, there were an estimated 431 288 new cases of kidney cancer (Renal Cell Carcinoma, RCC) globally with 138 611 cases in Europe, leading to 179 368 deaths worldwide, including 54 054 deaths in Europe (source: IARC/Globocan). To define high priority topics in academic research and launch dedicated trials, European RCC academic physicians have gathered into a European initiative - the CARE group.

Systemic therapy for RCC relies on two classes of agents: anti-angiogenic targeted therapy (Vascular endothelial growth factor Tyrosine Kinase Inhibitor- VEGFR TKI) and immune checkpoint inhibitor (ICI), targeting either PD-1/PD-L1 axis or CTLA-4. Combination therapy is standard of care (SOC) for clear cell RCC in all guidelines with either ICI-ICI or ICI-VEGFR TKI. However, no head-to-head comparison have been performed between the two approaches and patients are treated based on physician decision without clinical or biomarker factors to guide treatment selection. PD-L1 staining is, to date, the biomarker that has demonstrated its ability to enrich for overall survival benefit favoring ICI-ICI strategy in PD-L1(+) and ICI-VEGFR TKI in PD-L1(-) patients.

CARE1 PCT is a prospective randomize phase III study, in first line setting for patients with metastatic clear cell RCC comparing ICI-ICI vs ICI-VEGFR TKI approaches stratified on PD-L1 by local determination. Primary endpoint is overall survival (OS). The trial will enroll 1250 patients over 4 years across eight European countries (France, Spain, Netherlands, Czech Republic, Austria, Germany, Italy, UK) that are part of the CARE consortium. Study Sponsor is Gustave Roussy institute within the GETUG network for France, co-sponsor is developed through main academic networks (eg. SOGUG in Spain) and main institutions across Europe (eg. Cancer Core Europe - CCE). Study design has been develop to demonstrate that ICI-ICI is superior to ICI-VEGFR TKI in prolonging OS for PD-L1(+) patients and that ICI-VEGFR TKI is superior to ICI-ICI in prolonging OS for PD-L1(-) patients. CARE1 PCT has been designed and will be conducted with patient advocacy group representatives (ARTuR and IKCC) input.

CARE1 is an academic phase III study designed to define the optimal combination using a pragmatic routinely implementable biomarker. Therefore, CARE1 will inform practice and has the potential to change treatment guidelines. Taken all together, CARE1 is a unique opportunity to build a large-scale platform to define new biomarker based therapy guidelines as well as to investigate quality of life, patient reported outcome and Health-Economic in front line setting, as well as pathological and blood biobank collection for further translational work. This action is part of the Cancer Mission cluster of projects on 'Diagnosis and treatment'.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic (AJCC Stage IV) renal cell carcinoma with a clear-cell component.
2. Intermediate- or poor-risk mRCC as defined by IMDC classification.
3. Adult male or female patients (≥ 18 years of age at inclusion).
4. Karnofsky Performance Status (KPS) ≥70%.
5. Adequate organ and marrow function, according to investigator assessment and

   1. Absolute neutrophil count (ANC) ≥ 1000/μL (≥ 1.5 GI/L)
   2. Platelets ≥ 100,000/μL (≥ 100 GI/L)
   3. Hemoglobin ≥ 8 g/dL (≥ 80 g/L)
   4. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 x ULN.
   5. Calculated creatinine clearance ≥ 30 mL/min (≥ 0.67 mL/sec) using the CKD- EPI equation
6. Patient should understand, sign, and date the written informed consent form prior to any protocol-specific procedures performed.
7. Patient should be able and willing to comply with study visits and procedures as per protocol
8. Patients must be affiliated to a social security system or beneficiary of the same
9. Female patients must either be of non-reproductive potential or must have a negative serum pregnancy test within 14 days prior to the administration of study drug. Childbearing potential women must have agreed to use one barrier method of contraception, such as condom, plus an additional highly effective method of contraception during treatment on this trial and for up to 5 months after the last dose of study treatment.
10. Fertile men with a female partner of childbearing potential must agree to use one barrier method of contraception, such as condom, during treatment on this trial and for up to 4 months after the last dose of treatment. Their women of childbearing potential partner must agree to use a highly effective method of contraception during the same period.
11. Female subjects of childbearing potential must not be pregnant at screening.

Exclusion Criteria:

1. Prior systemic anticancer therapy for mRCC including investigational agents. Note: One prior systemic adjuvant therapy is allowed for completely resected RCC and if recurrence occurred at least 6 months after the last dose of adjuvant therapy.
2. Uncontrolled brain metastases (adequately treated with radiotherapy and/or radiosurgery prior to randomization are eligible). Subjects who are neurologically symptomatic as a result of their CNS metastasis or are receiving systemic corticosteroid treatment (prednisone equivalent > 10 mg/day) at the planned time of randomization are not eligible.
3. Concomitant oral anti-vitamin K anticoagulation. An exception is the use of LMWH or direct oral anticoagulants (DOAC), if considered safe by investigator assessment.
4. The subject has uncontrolled, significant intercurrent or recent illness such as the following conditions:

   a. Cardiovascular disorders:

   i. Congestive heart failure (CHF) class III or IV as defined by the New York Heart Association, unstable angina pectoris, myocardial infarction, serious cardiac arrhythmias (e.g., ventricular flutter, ventricular fibrillation, Torsades de pointes).

   ii. Uncontrolled hypertension despite optimal antihypertensive treatment.

   iii. Stroke, or other symptomatic ischemic event or severe thromboembolic event (e.g., symptomatic pulmonary embolism [PE], incidental PE is acceptable if deemed safe by the investigator) within 3 months before randomization.

   b. Active GI bleeding or symptomatic Gastrointestinal (GI) tract obstruction

   c. Clinically significant bleeding including uncontrolled hematuria, hematemesis, or hemoptysis

   d. Autoimmune disease that has been symptomatic or required immunosuppressive systemic treatment within the past two years from the date of randomization.

   Note: Patients with a history of Crohn's disease or ulcerative colitis are always excluded

   e. Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of randomization.

   Note: Inhaled, intranasal, intra-articular, or topical steroids are permitted. Adrenal replacement steroid doses > 10 mg daily prednisone equivalent are permitted. Transient short-term use of systemic corticosteroids for allergic conditions (e.g., contrast allergy) is also allowed.

   f. Active infection requiring systemic treatment.

   g. Major surgery (e.g., nephrectomy, GI surgery, removal of brain metastasis) within 4 weeks prior to randomization or serious non-healing wound/ulcer/bone fracture.
5. Pregnant or breastfeeding females.
6. Any other active malignancy at time of randomization or diagnosis of another malignancy within 3 years prior to randomization that requires active treatment, except for locally curable cancers that have been apparently cured.
7. Hypersensitivity to any of the active substances or to any of the excipients administered during the study
8. Use of live vaccines within 28 days before randomization
9. Persons deprived of their freedom or under guardianship, or for whom it would be impossible to undergo the medical follow-up required by the trial, for geographic, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1250 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2032-05-05 (Estimated); Study Completion 2032-05-05 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS). | At end of study, 97 months
  From randomization to time of death

SECONDARY OUTCOMES:
Progression-free survival according to RECIST 1.1 | At end of study, 97 months
  From randomization to progression, also a primary outcome for PDL1(-) population.
Objective Response Rate (ORR) according to RECIST 1.1 | At end of treatment, 60 months
  ORR (estimand 3) is defined as the percentage of randomised participants (ITT set) who achieve a best response of complete response (CR) or partial response (PR) over the treatment observation period based on Investigators assessments.
Quality of Life via questionnaire EQ-5D-5L | Baseline, Month 3, Month 6, Month 9, Month 12
  Patient's response to the Quality of Life questionnaire EQ-5D-5L.
Quality of Life via questionnaire NNCCN/FACT Kidney Cancer Symptom Index (NFKSI) | Baseline, Month 3, Month 6, Month 9, Month 12
  Patient's response to the Quality of Life questionnaire NFKSI19.
Quality of Life via questionnaire Kidney Symptom Index (KSI) | Baseline, Month 3, Month 6, Month 9, Month 12
  Patient's response to the Quality of Life questionnaire KSI.
Duration of Treatment | At end of treatment, 60 months
  Duration of protocolar treatment administration.
Time to treatment discontinuation (TTD) | At end of treatment, 60 months
  TTD is defined as the time from the date of treatment initiation to the date of last treatment dose.
Treatment-free survival (TFS) | At end of study, 97 months
  TFS is defined as the date from protocol therapy cessation (whatever the reason) to the date of subsequent systemic therapy initiation or death.
Time to subsequent systemic anticancer therapy (TTSST) | At end of study, 97 months
  TTSST is defined the time from the date of randomization to the date of next subsequent systemic therapy.
Incidence of AE's | At end of treatment, 60 months
  Incidence of AEs will be summarized by system organ class and preferred term according to MedDRA coding, and will be presented by treatment groups and overall.
Health Economic evaluation: healthcare costs [France & Netherlands only] | At end of study, 97 months
  The cost difference between arms in each patient subgroup (comparison of healthcare costs)
Health Economic evaluation: cost-utility [France & Netherlands only] | At end of study, 97 months
  The incremental cost per QALY and the incremental net monetary benefit in each patient subgroup (cost-utility analysis).

CONTACTS AND LOCATIONS:
Overall Officials: Laurence ALBIGES, MD, PhD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (46):
- Medical University of Vienna, Vienna, Austria
- Czechia (4):
  - Masarykův onkologický ústav, Masaryk Memorial Cancer Institute (MOU), Brno
  - Fakultní nemocnice Hradec Králová, University Hospital Hradec Kralove (FNHK), Hradec Králové
  - Fakultní nemocnice Olomouc, University Hospital Olomouc (FNOL), Olomouc
  - Fakultní nemocnice v Motole, University Hospital Motol (MOTOL), Prague
- France (40):
  - Institut de Cancérologie de l'Ouest - Angers, Angers
  - CHU Angers, Angers
  - Institut Sainte Catherine, Avignon
  - CH de la Côte Basque, Bayonne
  - Hôpital Jean Minjoz, Besançon
  - CHU de Bordeaux Hôpital Saint-André, Bordeaux
  - Centre François Baclesse, Caen
  - CH Châlon Sur Saône, Chalon-sur-Saône
  - Centre Jean Perrin, Clermont-Ferrand
  - Hôpital Henri Mondor, Créteil
  - Centre Georges-François Leclerc, Dijon
  - CHU Grenoble, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - Centre Oscar Lambret, Lille
  - Polyclinique de Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Institut Régional du Cancer de Montpellier, Montpellier
  - Centre Antoine Lacassagne, Nice
  - CHU de Nîmes, Nîmes
  - Hôpital de la Pitié Salpêtrière, Paris
  - Hôpital Bichat - Claude Bernard, Paris
  - Hôpital Tenon, Paris
  - Hôpital Saint-Louis, Paris
  - Institut Mutualiste Montsouris, Paris
  - CH de Pau, Pau
  - Hospices Civils de Lyon, Pierre-Bénite
  - CHU Poitiers, Poitiers
  - Institut Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - CHU Saint-Etienne, Saint-Etienne
  - Institut de Cancérologie de l'Ouest - Saint Herblain, Saint-Herblain
  - HIA Bégin, Saint-Mandé
  - CHU Sud Réunion, Saint-Pierre
  - Institut de cancérologie Strasbourg Europe, Strasbourg
  - Hôpital Foch, Suresnes
  - Oncopole Claudius Regaud - IUCT-Oncopole, Toulouse
  - Hôpital Bretonneau, Tours
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif
- Antoni van Leeuwenhoek, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No